CLINICAL TRIAL: NCT00276679
Title: Phase II Study of Temozolomide (Temodal) in Children Over 1 Year of Age With Relapsed or Refractory High Risk Neuroblastoma
Brief Title: Temozolomide in Treating Young Patients With High-Risk Relapsed or Refractory Neuroblastoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Non-Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454577; CCLG-NAG-2003-02; EU-20591; CCLG-SFOP-NAG-2003-02
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2006-01

CONDITIONS: Neuroblastoma
Keywords: recurrent neuroblastoma; disseminated neuroblastoma; localized unresectable neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — Temozolomide

INTERVENTIONS:
Drug: temozolomide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well temozolomide works in treating patients with high-risk relapsed or refractory neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the anti-tumor activity of temozolomide in young patients with high-risk relapsed or refractory neuroblastoma.

Secondary

* Determine the duration of response in patients treated with this drug.
* Determine tolerability of this drug in these patients
* Determine the tumor expression of the cellular repair mechanisms which repair DNA damage (O6-methylguanine-DNA methyltransferase [MGMT] and mismatch repair [MMR] systems) in patients treated with this drug.
* Correlate MGMT and MMR expression with outcomes in patients treated with this drug.
* Determine if MGMT and MMR expression/activity changes in the tumor during initial presentation, treatment, and relapse/progression in patients treated with this drug.
* Determine the activity of MGMT in bone marrow taken at relapse, in terms of hematological toxicity, in patients treated with this drug.

OUTLINE: This is a multicenter, open label, nonrandomized study.

Patients receive oral temozolomide once daily for 5 days. Treatment repeats every 28 days for 2 courses. Patients achieving stable or responding disease after completion of the 2 courses may receive up to 10 additional courses of treatment in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven neuroblastoma

  * High-risk relapsed or refractory disease, defined as 1 of the following:

    * Metastatic disease
    * Localized MYC-N amplified disease
    * Localized non MYC-N amplified disease at second relapse
* Measurable primary or metastatic disease by cross-sectional imaging or MIBG scan

PATIENT CHARACTERISTICS:

* Lansky performance status 40-100%
* Life expectancy > 2 months
* Not pregnant or nursing
* Fertile patients must use effective contraception during the course of this study and for 6 months after study completion
* Organ toxicity < grade 2
* Platelets ≥ 100,000/mm^3 (50,000/mm^3 after stem cell transplant or in case of marrow involvement)
* Neutrophil count ≥ 500/mm^3
* Bilirubin < 1.5 times normal
* AST and ALT ≤ 2.5 times normal
* No known HIV positivity

PRIOR CONCURRENT THERAPY:

* More than 21 days since prior chemotherapy treatment (isotretinoin is counted as chemotherapy for this purpose)
* More than 30 days since prior radiotherapy except local palliative treatment for pain control
* No more than 2 prior treatments for neuroblastoma
* No other concurrent investigative treatment for neuroblastoma

Ages: 1 Year to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-04; Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herve Rubie, MD, Study Chair — Centre Hospitalier Regional de Purpan; Andrew David J. Pearson, MD, FRCP, DCh — University of Newcastle Upon-Tyne; Julia Chisholm, MD — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (22):
- Centre Hospitalier Regional de Purpan, Toulouse, France
- Our Lady's Hospital for Sick Children, Dublin, Ireland
- United Kingdom (20):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital at Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children NHS Trust, London, England
  - Central Manchester and Manchester Children's University Hospitals NHS Trust, Manchester, England
  - Sir James Spence Institute of Child Health, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden NHS Foundation Trust - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales

REFERENCES:
- [Result] Rubie H, Chisholm J, Defachelles AS, Morland B, Munzer C, Valteau-Couanet D, Mosseri V, Bergeron C, Weston C, Coze C, Auvrignon A, Djafari L, Hobson R, Baunin C, Dickinson F, Brisse H, McHugh K, Biassoni L, Giammarile F, Vassal G; Societe Francaisedes Cancers de l'Enfant; United Kingdom Children Cancer Study Group-New Agents Group Study. Phase II study of temozolomide in relapsed or refractory high-risk neuroblastoma: a joint Societe Francaise des Cancers de l'Enfant and United Kingdom Children Cancer Study Group-New Agents Group Study. J Clin Oncol. 2006 Nov 20;24(33):5259-64. doi: 10.1200/JCO.2006.06.1572. PMID 17114659